CLINICAL TRIAL: NCT03536143
Title: A Phase I/II Study of KB103, a Non-Integrating, Replication-Incompetent HSV Vector Expressing the Human Collagen VII Protein, for the Treatment of Dystrophic Epidermolysis Bullosa (DEB)
Brief Title: A Phase I/II Study of KB103, a Topical HSV1-COL7, on DEB Patients
Acronym: GEM-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB103-001
Record Dates: First submitted 2018-04-20; First posted 2018-05-24 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-11

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: bullosa; DEB; RDEB; Krystal; epidermolysis; Beremagene; Geperpavec; KB103; HSV-COL7A1
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: Intrasubject treatment assignment/randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical beremagene geperpavec (Experimental): HSV1-COL7A1 vector (KB103)
  Interventions: Biological: Topical beremagene geperpavec
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo gel

INTERVENTIONS:
Biological: Topical beremagene geperpavec — Topical gel of non-integrating, replication-incompetent HSV-1 expressing the human collagen VII protein
  Other Names: HSV1-COL7A1; KB103
  Arms: Topical beremagene geperpavec
Biological: Placebo gel — Placebo gel
  Arms: Placebo

SUMMARY:
This study was conducted to assess the safety and efficacy of topical Beremagene Geperpavec (KB103, HSV1-COL7) on DEB patients.

DETAILED DESCRIPTION:
The primary objectives were the evaluation of safety, through incidence of adverse events associated with the administration of B-VEC as compared to placebo, as well as the demonstration of molecular correction of the disease by establishing the presence of functional COL7 expression and anchoring fibrils (AF) formation post administration of B-VEC. Additional primary objectives were to assess the proportion of wounds with complete wound closure (≥90% reduction from baseline wound surface area) at Week 8, 10, and 12, the duration of wound closure, and the time to wound closure of B-VEC treated wounds as compared with placebo treated wounds.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the recessive form of dystrophic epidermolysis bullosa (RDEB).
* Age

  1. Phase 1: 18 years old or older,
  2. Phase 2a: 5 years old or older,
  3. Phase 2b: 2 years old or older,
  4. Phase 2c: 2 years old or older.
* Willing and able to give consent/assent
* Confirmation of RDEB diagnosis by genetic testing, IF, and IEM
* LH24 antibody negative (non-collagenous [NC] 2domain [NC2-]) and NC1 domain [NC1+]). (This criterion is applicable to the first 2 adults on the study (Phase 1). Subsequent subjects can be NC1+ or NC1-)
* Confirmed RDEB COL7A1 mutations in subject
* Wound that meets the wound size/surface area entry criteria:

  1. Phase 1: Two wounds up to 10 cm2; 1 randomized to B-VEC and 1 randomized to placebo
  2. Phase 2a and 2b: At least 3 wounds up to 20 cm2; 2 wounds randomized to B-VEC and 1 randomized to placebo
  3. Phase 2c: At least 2 wounds up to 50 cm2; at least 1 randomized to B-VEC and 1 randomized to placebo
* Subjects, who are, in the opinion of the investigator, able to understand the study, cooperate with the study procedures, and are willing to return to the clinic for all the required follow-up visits.

Exclusion Criteria:

* Medical instability limiting ability to travel to the investigative center
* The presence of medical illness expected to complicate participation and/or compromise the safety of this technique, such as active infection with human immunodeficiency virus (HIV), hepatitis B (as determined by hepatitis B surface antigen screening), or hepatitis C (as determined by detection of hepatitis C antibodies, or positive result of hepatitis C polymerase chain reaction [PCR] analysis)
* Serum antibodies to COL7 demonstrated on enzyme-linked immunosorbent assay (ELISA), indirect immunofluorescence microscopy, Western blot, or cell-mediated immunity to enzyme-lined ImmunoSpot® (subjects with negative results within 12 months of screening are eligible)
* Active infection in the area that will undergo administration
* Evidence of systemic infection
* Known allergy to any of the constituents of the product
* Current evidence or a history of squamous cell carcinoma in the area that will undergo treatment
* Active drug or alcohol addiction
* Hypersensitivity to local anesthesia (lidocaine/prilocaine cream)
* Receipt of chemical or biological study product for the specific treatment of RDEB in the past 3 months
* Specific wounds that have previously been administered investigational gene or cell therapy
* Subjects who have taken systemic antibiotics within 7 days
* Positive pregnancy test or breast-feeding
* Clinically significant abnormalities as determined by the investigator

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gurevich I, Agarwal P, Zhang P, Dolorito JA, Oliver S, Liu H, Reitze N, Sarma N, Bagci IS, Sridhar K, Kakarla V, Yenamandra VK, O'Malley M, Prisco M, Tufa SF, Keene DR, South AP, Krishnan SM, Marinkovich MP. In vivo topical gene therapy for recessive dystrophic epidermolysis bullosa: a phase 1 and 2 trial. Nat Med. 2022 Apr;28(4):780-788. doi: 10.1038/s41591-022-01737-y. Epub 2022 Mar 28. PMID 35347281

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Wounds
Groups:
- All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo"): The randomization scheme and subject-specific randomization envelopes were created for each phase of the study for each subject. At the baseline visit, subjects were assigned a randomization number and the investigator selected either 2 (Phase 1, B-VEC: Placebo = 1:1), 3 (Phase 2a and 2b, B-VEC: Placebo = 2:1), or 2 (Phase 2c, B-VEC: Placebo = 1:1) similar sized wounds, as applicable. Using the randomization scheme with the subject-specific envelope, the wounds were assigned to either B-VEC or placebo.
Period: Overall Study
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
Started | 12; 33 Wounds (The numbers of wounds selected for each subject were 2 in Phase 1 (2 subjects, B-VEC: Placebo = 1:1), 3 in Phase 2a and 2b (9 subjects, B-VEC: Placebo = 2:1), and 2 in Phase 2c (1 subject, B-VEC: Placebo = 1:1). The total wounds selected for this study were 33 (=2x2+9x3+2x1), in which 21 received B-VEC and 12 received Placebo.)
B-VEC | 12; 21 Wounds
Placebo | 12; 12 Wounds
Completed | 11; 31 Wounds
Not Completed | 1; 2 Wounds
Not completed — Early termination, Sponsor decision | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo"): The randomization scheme and subject-specific randomization envelopes were created for each phase of the study. At the baseline visit, subjects were assigned a randomization number and the investigator selected either 2 (Phase 1, B-VEC: Placebo = 1:1), 3 (Phase 2a and 2b, B-VEC: Placebo = 2:1), or 2 (Phase 2c, B-VEC: Placebo = 1:1) similar sized wounds, as applicable. Using the randomization scheme with the subject-specific envelope, the wounds were assigned to either B-VEC or placebo.
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.3 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race : White | 12
  Ethnicity : Hispanic or Latino | 3
  Ethnicity : Not Hispanic or Latino | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reported at Least One Adverse Event, Safety Population
Description: Safety assessments included evaluation of medical and medication history, physical / skin examination, vital signs, adverse events, and laboratory evaluations. Due to the 'split-person' intrasubject design, the safety assessments were reported at subject level, but not per intervention.
Time Frame: baseline to 12 weeks
Population: Safety population included all subjects administered B-VEC or Placebo. Due to the 'split-person' intrasubject design, the safety assessments were reported at subject level, but not per intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
Number analyzed (Participants) | 12
Participants | 9

2. Primary Outcome: Number of Adverse Events Reported, Safety Population
Description: as for outcome 1
Time Frame: baseline to 12 weeks
Population: as for outcome 1
Measure: Number; unit: number of adverse events
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
Number analyzed (Participants) | 9
number of adverse events | 35

3. Primary Outcome: Complete Wound Closure Responder, ITT Population
Description: One wound is a responder if the reduction from baseline in wound surface is ≥90%.
Time Frame: from baseline at Weeks 8, 10, and 12
Population: The intent-to-treat (ITT) population: subjects who were administered KB103 who have had at least one paired assessment of the target wound area post-administration, i.e., at least one KB103 target wound and one placebo target wound.
  The Safety population: all subjects who were administered IP. The per-protocol (PP) population: all subjects in the ITT population who have had at least one paired assessment of the target wound area post-administration and completed the protocol as planned.
Measure: Number; unit: number of responder
Units Other Than Participants: Wounds
Groups:
- B-VEC: The wounds assigned to B-VEC.
- Placebo: The wounds assigned to Placebo.
Arm/Group | B-VEC | Placebo
Number analyzed (Participants) | 11 | 11
Number analyzed (Wounds) | 20 | 11
number of responder
  Week 8: number analyzed (Wounds) | 17 | 8
  Week 8 | 14 | 0
  Week 10: number analyzed (Wounds) | 16 | 6
  Week 10 | 12 | 2
  Week 12: number analyzed (Wounds) | 14 | 7
  Week 12 | 12 | 1

4. Primary Outcome: Time to Wound Closure Analysis, ITT Population
Description: Time to wound closure was defined as the time from the first treatment to Complete Wound Closure (≥90% reduction in wound surface area from baseline)
Time Frame: baseline to complete wound closure
Population: Intent to treat (ITT) included all subjects who were administered IP and had at least 1 post dose paired wound assessment.
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Wounds
Groups:
- Placebo: Placebo
  Topical beremagene geperpavec: Topical gel of non-integrating, replication-incompetent HSV-1 expressing the human collagen VII protein
Arm/Group | Topical Beremagene Geperpavec | Placebo
Number analyzed (Participants) | 11 | 11
Number analyzed (Wounds) | 20 | 11
days | 13.5 [8.0 to 21.0] | 22.5 [8.0 to 64.0]
Statistical Analysis 1: Comparison: Topical Beremagene Geperpavec vs Placebo; Test type: Superiority; p = 0.0216, Log Rank

5. Primary Outcome: Duration of Wound Closure, ITT Population
Description: Duration of wound closure
Time Frame: Time from the complete closure to the first reopening of the same wound
Population: ITT population included all subjects who were administered IP and had at least 1 post dose paired wound assessment.
Measure: Median (95% Confidence Interval); unit: days
Units Other Than Participants: Wounds
Arm/Group | Topical Beremagene Geperpavec | Placebo
Number analyzed (Participants) | 11 | 11
Number analyzed (Wounds) | 20 | 11
days | 103.0 [94.0 to 118.0] | 16.5 [0.0 to 66.0]
Statistical Analysis 1: Comparison: Topical Beremagene Geperpavec vs Placebo; Test type: Superiority; p = 0.0009, Log Rank

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo"): The randomization scheme and subject-specific randomization envelopes were created for each phase of the study. At the baseline visit, subjects were assigned a randomization number and the investigator selected either 2 (Phase 1, B-VEC: Placebo = 1:1), 3 (Phase 2a and 2b, B-VEC: Placebo = 2:1), or 2 (Phase 2c, B-VEC: Placebo = 1:1) similar sized wounds, as applicable. Using the randomization scheme with the subject-specific envelope, the wounds were assigned to either B-VEC or placebo.
  Due to the 'split-person'/intrasubject design, each subject received both B-VEC and Placebo. Therefore, the safety assessments were reported at subject level, but not per intervention. The site/treatment specific information on AEs was not systematically collected in a prospective fashion, therefore it was not reported.
Arm/Group | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo")
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants ("Topical Beremagene Geperpavec (B-VEC)", and "Placebo") (N=12)
Application site pruritus (General disorders) | 2 (2)
Application site bruise (General disorders) | 1 (1)
Application site erythema (General disorders) | 1 (1)
Application site rash (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (2)
Injection site pain (General disorders) | 1 (3)
Injection site swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Purulent discharge (Infections and infestations) | 1 (2)
Wound infection pseuomonas (Infections and infestations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Bacterial test positive (Investigations) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 1 (1)
Wound Treatment (Surgical and medical procedures) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Product taste abnormal (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT03536143/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03536143/SAP_001.pdf